CLINICAL TRIAL: NCT04791709
Title: Preventing Cognitive Decline in HIV-infected Latinos Through a Culturally Tailored Health Promotion Intervention (HOLA)
Brief Title: Happy Older Latinos Are Active - Cognitive Decline
Acronym: HOLA-CD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Daniel Enrique Jimenez, Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20201202; U54MD002266-14S1 (NIH)
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HOLA Group (Experimental): Participants in this group will receive a multicomponent intervention for 16 weeks.
  Interventions: Behavioral: Happy Older Latinos are Active (HOLA)

INTERVENTIONS:
Behavioral: Happy Older Latinos are Active (HOLA) — HOLA is a multicomponent health promotion intervention. First component is a one-on-one social and physical activation with the participant and the community health worker (CHW). Each session will last approximately 30 minutes at day 1 and week 8. The second component is a group walk led by a CHW for 45 minutes, 3 times a week, for 16 weeks. The third component consists of scheduling pleasant events at the end of each group walk session.

SUMMARY:
The purpose of this study is to look at the best ways to prevent cognitive decline (loss of memory and/or functioning) in midlife and older Latino adults living with HIV.

DETAILED DESCRIPTION:
The purpose of this study is to look at the best ways to prevent cognitive decline (loss of memory and/or functioning) in midlife and older Latino adults living with HIV. It assesses the feasibility of running a health promotion program, led by a community health worker (CHW) intended to help prevent cognitive decline (loss of memory and/or functioning) through a culturally tailored health promotion intervention . Eligible participants will be Latino/Hispanic individuals 50 years of age or older, living with HIV, who may be at risk of developing chronic diseases such as dementia and Alzherimer's.

ELIGIBILITY:
Inclusion Criteria:

* are Latino (self-identified);
* are age 50+;
* are HIV infected but are virologically suppressed (viral load <200 copies/mL);
* volunteer informed consent

Exclusion Criteria:

* have diagnosis of any neurodegenerative disorder or dementia (Parkinson's disease, Alzheimer's disease, vascular, frontotemporal dementia, etc.) or significant cognitive impairment as indicated by a Telephone Interview for Cognitive Status (TICS) score less than or equal to 30;
* have other conditions that could impact cognitive functioning or testing (e.g., legally blind or deaf), currently undergoing radiation or chemotherapy, a history of brain trauma with a loss of consciousness greater than 30 minutes.
* have contraindications to physical activity outlined in the American College of Sports Medicine standards or severe medical illness that precludes them from safely participating in a health promotion intervention.
* are unable to complete 10-meter walk test.
* have plans to move outside of the Miami metropolitan area within the next 6 months or are not living in stable housing (e.g. group home).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Jimenez, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jimenez DE, Ross EJ, Weinstein E, Gouse H, Pan Y, Martinez Garza D, Burke SL, Joo JH, Behar-Zusman V. Preventing Cognitive Decline in Older Latino Adults With HIV Through a Culturally Tailored Health Promotion Intervention: Protocol for a Single-Arm Pilot Trial. JMIR Res Protoc. 2024 Aug 12;13:e55507. doi: 10.2196/55507. PMID 39133532

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HOLA Group
Started | 30
Completed | 27
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | HOLA Group
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 25
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Completing the Study
Description: Feasibility of HOLA will be reported as the percentage of participants completing the post intervention assessment.
Time Frame: 16 weeks
Measure: Number; unit: Percentage of participants
Arm/Group | HOLA Group
Number analyzed (Participants) | 30
Percentage of participants | 90

2. Secondary Outcome: Changes in Neurocognitive Impairment as Measured by the Trails Making Test
Description: Trail Making Test (TMT). Time to accurately complete Part A and Part B. The TMT measures neurocognitive functioning and consists of two parts; the first part requires participants to connect numbers in ascending order, while the second part requires individuals to connect numbers and letters in sequence. The test is scored by the time it takes to accurately complete each test. Increases in time correlate with greater impairment measured in seconds.
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | HOLA Group
Number analyzed (Participants) | 27
seconds
  Trail Making Test (TMT) A-Baseline | 48.7 (24.0)
  Trail Making Test (TMT) B-Baseline | 172.0 (79.0)
  Trail Making Test (TMT) A-16 weeks | 44.3 (19.0)
  Trail Making Test (TMT) B-16 weeks | 137.0 (70.6)

3. Secondary Outcome: Changes in Neurocognitive Impairment as Measured by the WAIS-IV Digit Span
Description: The Wechsler Adult Intelligence Scale-Fourth Edition (WAIS-IV) asks participants to repeat 2-9 numbers forward, backward and in ascending order to assess attention, processing speed, and working memory. Each correct response earns 1 point, and the total raw score is converted to a scaled score ranging from 1 to 19. Higher scores indicate better cognitive performance; lower scores reflect increased neurocognitive impairment.
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HOLA Group
Number analyzed (Participants) | 27
score on a scale
  Baseline | 6.5 (1.93)
  16 weeks | 6.81 (2.34)

4. Secondary Outcome: Changes in Physical Activity as Measured by the Global Physical Activity Questionnaire (GPAQ)
Description: The Global Physical Activity Questionnaire (GPAQ) scoring is based on the amount of time a person spends being physically active in a typical week. It looks at three areas: activity at work or during daily tasks (including heavy lifting, digging, carrying loads, or light activities like cleaning); traveling from place to place (like walking or cycling); and recreational activities (such as exercise, sports, or active hobbies). Each activity is converted into a standard unit called MET-minutes (Metabolic Equivalent of Task). This allows different types of activity to be compared on the same scale. The total MET-minutes per week are calculated by multiplying: Minutes per day × Days per week × MET value with higher scores indicating greater levels of activity.
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: MET-minutes per week
Arm/Group | HOLA Group
Number analyzed (Participants) | 27
MET-minutes per week
  Baseline | 1,743 (2,842)
  16 weeks | 4,533 (5,008)

5. Secondary Outcome: Changes in Depression as Measured by the PHQ-9
Description: The Patient Health Questionnaire (PHQ-9) is a 9 item questionnaire that measures depression severity. The total score ranges from 0-27 with higher scores indicating more severe depression.
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HOLA Group
Number analyzed (Participants) | 27
score on a scale
  Baseline | 6.67 (4.84)
  16 weeks | 4.26 (3.35)

6. Secondary Outcome: Changes in Anxiety as Measured by the GAD-7
Description: The Generalized Anxiety Disorder (GAD-7) is a 7 item questionnaire that measures anxiety severity. The total score ranges from 0-21 with higher scores indicating more severe anxiety.
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HOLA Group
Number analyzed (Participants) | 27
score on a scale
  Baseline | 4.83 (3.97)
  16 weeks | 3.56 (2.81)

7. Secondary Outcome: Changes in Psychosocial Functioning as Measured by the MSPSS
Description: The Multidimensional Scale of Perceived Social Support (MSPSS) is a 12 item questionnaire that measures perceived social support. The total score ranges from 1-84 with higher scores indicating more perceived social support.
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HOLA Group
Number analyzed (Participants) | 27
score on a scale
  Multidimensional Scale of Perceived Social Support (MSPSS) baseline | 5 (1.2)
  Multidimensional Scale of Perceived Social Support (MSPSS) 16 weeks | 5 (1.2)

8. Secondary Outcome: Changes in Biomarkers of Cognition
Description: Biomarkers of cognition including interleukin-15, brain derived neurotrophic factor (BDNF), and vascular endothelial growth factor (VEG-F) reported in pg/ml will be assessed from blood samples.
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | HOLA Group
Number analyzed (Participants) | 27
pg/ml
  interleukin-15 Baseline | 6.6 (1.26)
  interleukin-15 16 weeks | 6.6 (1.5)
  brain derived neurotrophic factor (BDNF) baseline | 3117.1 (1853.5)
  brain derived neurotrophic factor (BDNF) 16 weeks | 3411.3 (2336.5)
  vascular endothelial growth factor (VEG-F) baseline | 34.1 (22.1)
  vascular endothelial growth factor (VEG-F) 16 weeks | 32.3 (18.1)

9. Secondary Outcome: Changes in Biomarkers of Cognition Levels
Description: Biomarkers of cognition levels including irisin and insulin like growth factor (IGF-1) reported in ng/ml will be assessed from blood samples.
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | HOLA Group
Number analyzed (Participants) | 27
ng/ml
  irisin Baseline | 39.9 (36.1)
  irisin 16 weeks | 36.6 (30.8)
  insulin like growth factor (IGF-1) baseline | 79.4 (51.1)
  insulin like growth factor (IGF-1) 16 weeks | 65.8 (34.3)

10. Secondary Outcome: Changes in Adiponectin
Description: Adiponectin will be assessed from blood samples measured by ng/ml
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | HOLA Group
Number analyzed (Participants) | 27
ng/ml
  Baseline | 13999.1 (3571.6)
  16 weeks | 14289.6 (3946.8)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | HOLA Group
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT04791709/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/09/NCT04791709/ICF_001.pdf